CLINICAL TRIAL: NCT06789731
Title: Mindfulness-Based Interventions Targeting First-Generation College Student Retention in Rural Environments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-117
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either: 1) Mindfulness Meditation or 2) Psychoeducation
Who Masked: Outcomes Assessor
Masking Description: The PI will randomly assign participants to condition and coordinate treatment group scheduling; the assessor will be blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation (Experimental): Participants will meet virtually with the mindfulness practitioner once a week for four weeks for 30-minute segments.
  Interventions: Behavioral: Mindfulness Meditation
- Psychoeducation (Active Comparator): Participants will receive recordings online, once a week for four weeks which will be approximately 30 minutes in length.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness Meditation — Mindfulness meditation will be facilitated by a seasoned mindfulness practitioner. Participants will be guided through a loving kindness meditation adapted to apply to college communities and designed to help increase a sense of interconnectedness among their college community. They will also learn how to deconstruct feelings of anxiety and/or depression into sensory, emotional, cognitive, and behavioral components.
  Arms: Mindfulness Meditation
Other: Psychoeducation — In the psychoeducation arm, participants will receive information related to creating connections with campus community and managing anxiety and/or depression through a presentation. They will also receive information on resources for connecting with their community and treating anxiety and/or depression.
  Arms: Psychoeducation

SUMMARY:
The goal of this randomized control group is to learn about effective treatments for college students experiencing anxiety and/or depression. The main questions this clinical trial aims to answer are: 1) Can mindfulness-based treatments increase retention rates among first-generation college students? 1) Can mindfulness-based treatments decrease anxiety and/or depression among first-generation college students?

Participants will be randomly assigned to one of two intervention groups: mindfulness meditation or psychoeducation. Researchers will compare outcomes from each group to explore treatment differences.

DETAILED DESCRIPTION:
Method/Design. This study will be a remote, two-arm, randomized, controlled trial. First-generation college students (N=53) will be randomized to either mindfulness meditation (MM), or psychoeducation (PE). The mindfulness meditation will be a loving kindness meditation adapted to apply to college communities. Each intervention will be applied for 30 minutes, once a week, for four weeks through a remote platform. The MM is adapted through a validated brief mindfulness-based intervention framework (Zeidan, 2010). The primary outcome, intention to persist in college, and the secondary outcomes, depression and anxiety, will be assessed by a blinded researcher at baseline, one-week post treatment, and one-month follow-up. Change in sense of connection during the final treatment session, measured with a comprehensive battery of self-report indices, will be the primary therapeutic mechanism.

Aims and Objectives. The proposed project's central hypothesis is that MM will increase first-generation students' intention to persist in college and increase their emotional well-being by increasing their sense of belonging in their college community. Aim 1. Examine MM's effect on first-generation college students' intention to persist in college (primary outcome) over time. Hypothesis: Participants who are randomized into the MM group will report higher intention to persist scores from baseline to one-month follow-up than those who are randomized to PE. Aim 2.

Exploratory. Determine MM's effect on anxiety and depression scores (co-secondary outcomes) over time. Hypothesis: MM will decrease depression and anxiety relative to PE from baseline to one-month follow-up. Aim 3: Exploratory. Investigate whether transcendent states during the final MM session predicts students' intention to persist scores. Hypothesis: The effect of MM on students' intention to persist will be mediated by self-transcendent experience during mindfulness practice.

ELIGIBILITY:
Inclusion Criteria:

18 years or older. Currently enrolled in four-year college in the United States. First-generation college student. Access to WiFi and a computer/smartphone/tablet. English speaking.

Exclusion Criteria:

Not currently enrolled in a four-year college. Not a first-generation college student. Non-English speaker. Not able to utilize WiFi or computer/tablet/smartphone.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Intention to Persist in College | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session)
  Change in participants' intention to persist in college will be assessed through an individual item rated in a numeric rating scale. Scores range from 0 to 5 with higher scores reflecting greater intent to remain in college.

SECONDARY OUTCOMES:
Anxiety | Changes in participant's state anxiety will be captured within 5-minutes prior to each intervention and within 5 minutes after each intervention (mindfulness and psychoeducation)
  Symptoms will be assessed through a state anxiety assessment. Scores range from 0-60 with higher scores indicating higher levels of anxiety.
Depression | Changes in participant's state anxiety will be captured within 5-minutes prior to each intervention and within 5 minutes after each intervention (mindfulness and psychoeducation)
  Symptoms will be assessed through a state depression assessment. Scores range from 0-20 with higher scores indicating higher levels of depression.

OTHER OUTCOMES:
Adverse Childhood Experiences questionnaire | Baseline
  Participants adverse childhood experiences will be assessed at baseline to explore how childhood adversities moderate outcomes.The ACEs questionnaire was adapted from the Felitti et al., (1998) wave two survey and current questions used by the CDC's telephone Behavioral Risk Factor Surveillance System survey collected in all 50 states. ACES range between 0-13 and the higher the score, the higher the number of ACES.
Sensation Manikin | Changes in participant's state body sensations will be captured within 5-minutes prior to each intervention and within 5 minutes after each intervention (mindfulness, external qigong, and psychoeducation)
  Change in the distribution of pleasant and unpleasant bodily sensations. Scores can range from 0-100 for pleasant (higher scores indicate higher pleasant feelings) and 0-100 for unpleasant feelings (higher scores indicate higher levels of unpleasant sensations).
Perceived Discrimination | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session)
  Changes in the perception of experiencing discrimination (Everyday Discrimination). Scores range from 0 -54 with higher scores indicating higher levels of discrimination.
Connectedness to Nature Questionnaire | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session)
  The effects on Connectedness to Nature as a moderator between treatment and outcomes. The scale consists of 16 items rated on a 5-point Likert scale, from 1 (strongly disagree) to 5 (strongly agree) and is scored by creating a mean of the 16 items, with scores ranging from one to five, with higher scores indicating a stronger connectedness to nature than lower scores.
Dispositional Mindfulness Scale | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session)
  The Metacognitive Processes of Decentering scale (MPoD-t) will be used to assess the effects of dispositional mindfulness as a moderator between treatment and outcomes. Scores range from 0-80 with higher scores indicating higher dispositional mindfulness.
Sense of Belonging in College | Baseline, post treatment (one week after the final treatment session), and follow-up (one month after the final treatment session)
  The role of treatment type on the participant's sense of belonging in college. Scores range from 0-56 with higher scores indicating higher levels of belonging.
Trait Self-Transcendence | Changes in participant's self-transcendence will be captured within 5-minutes prior to each intervention and within 5 minutes after each intervention (mindfulness, external qigong, and psychoeducation)
  Change in self-transcendent state will be measured with the Nondual Awareness Dimensional Assessment - State Version. Scores range from 0 to 10, with higher scores reflecting greater self-transcendence.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Lecy, Principal Investigator — University of South Dakota
Locations (1):
- University of South Dakota, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steer RA, Brown GK, Beck AT, Sanderson WC. Mean Beck Depression Inventory-II scores by severity of major depressive episode. Psychol Rep. 2001 Jun;88(3 Pt 2):1075-6. doi: 10.2466/pr0.2001.88.3c.1075. PMID 11597055
- [Background] Hanley AW, Garland EL. Mapping the Affective Dimension of Embodiment With the Sensation Manikin: Validation Among Chronic Pain Patients and Modification by Mindfulness-Oriented Recovery Enhancement. Psychosom Med. 2019 Sep;81(7):612-621. doi: 10.1097/PSY.0000000000000725. PMID 31246748
- [Background] Hanley AW, Nakamura Y, Garland EL. The Nondual Awareness Dimensional Assessment (NADA): New tools to assess nondual traits and states of consciousness occurring within and beyond the context of meditation. Psychol Assess. 2018 Dec;30(12):1625-1639. doi: 10.1037/pas0000615. Epub 2018 Jul 30. PMID 30058824
- [Background] Knowles KA, Olatunji BO. Specificity of trait anxiety in anxiety and depression: Meta-analysis of the State-Trait Anxiety Inventory. Clin Psychol Rev. 2020 Dec;82:101928. doi: 10.1016/j.cpr.2020.101928. Epub 2020 Oct 10. PMID 33091745
- [Background] Sims M, Wyatt SB, Gutierrez ML, Taylor HA, Williams DR. Development and psychometric testing of a multidimensional instrument of perceived discrimination among African Americans in the Jackson Heart Study. Ethn Dis. 2009 Winter;19(1):56-64. PMID 19341164
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Navarro O, Olivos P, Fleury-Bahi G. "Connectedness to Nature Scale": Validity and Reliability in the French Context. Front Psychol. 2017 Dec 12;8:2180. doi: 10.3389/fpsyg.2017.02180. eCollection 2017. PMID 29312052